CLINICAL TRIAL: NCT03653338
Title: T-Cell Depleted, Alternative Donor Transplant in Pediatric and Adult Patients With Severe Sickle Cell Disease (SCD) and Other Transfusion-Dependent Anemias
Brief Title: T-Cell Depleted Alternative Donor Bone Marrow Transplant for Sickle Cell Disease (SCD) and Other Anemias
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Paul Szabolcs (Other)
Responsible Party: Sponsor-Investigator, Paul Szabolcs, Chief, Division of Blood and Marrow Transplantation and Cellular Therapy, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY19050050
Record Dates: First submitted 2018-08-02; First posted 2018-08-31 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Sickle Cell Anemia; Beta-thalassemia Major; Diamond-blackfan Anemia
Keywords: Sickle Cell; Diamond-Blackfan; Beta-thalassemia; Anemia; Stem cell transplantation; Unrelated Donor; haploidentical; hematopoietic stem cell transplant (HSCT); bone marrow transplant (BMT); mismatched; t-cell depletion
MeSH Terms: conditions — Anemia, Sickle Cell; beta-Thalassemia; Anemia, Diamond-Blackfan; Anemia | interventions — Hydroxyurea; Rituximab; Alemtuzumab; fludarabine; fludarabine phosphate; Thiotepa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Hematopoietic Stem Cell Transplantation (Experimental): All patients will receive a CD3+/CD19+ depleted stem cell transplant. In this study, the investigators will use HLA mismatched unrelated or haploidentical related donor peripheral blood stem cells. Prior to transplantation, the marrow (90-95%) will be negatively selected for CD3/CD19 using the ClinicMACs® depletion device. The remaining (5-10%) will undergo CD45+RA+ depletion and be frozen for future use as an immune boost.
  Subjects will undergo hematopoietic stem cell transplant utilizing CD3+/CD19+ depleted cells following conditioning therapy.
  Interventions: Biological: CD3/CD19 depleted leukocytes; Biological: CD45RA depleted leukocytes; Drug: Hydroxyurea; Drug: Rituximab; Drug: Alemtuzumab; Drug: Fludarabine; Drug: Thiotepa

INTERVENTIONS:
Biological: CD3/CD19 depleted leukocytes — Negative selection for CD3+/CD19+ cells will be performed on the CliniMACS® depletion device.
Biological: CD45RA depleted leukocytes — Negative selection for CD45RA will be performed on the CliniMACS® depletion device.
Drug: Hydroxyurea — Sickle Cell Disease Conditioning
  Other Names: HU, Hydrea
Drug: Rituximab — Sickle Cell Disease Conditioning
  Other Names: Rituxan
Drug: Alemtuzumab — Sickle Cell Disease Conditioning
  Other Names: Campath-1H
Drug: Fludarabine — Sickle Cell Disease Conditioning
  Other Names: Fludara
Drug: Thiotepa — Sickle Cell Disease Conditioning

SUMMARY:
The purpose of this study is to evaluate what effect, if any, mismatched unrelated volunteer donor and/or haploidentical related donor stem cell transplant may have on severe sickle cell disease and other transfusion dependent anemias. By using mismatched unrelated volunteer donor and/or haploidentical related donor stem cells, this study will increase the number of patients who can undergo a stem cell transplant for their specified disease. Additionally, using a T-cell depleted approach should reduce the incidence of graft-versus-host disease which would otherwise be increased in a mismatched transplant setting.

DETAILED DESCRIPTION:
CD3/CD19 depletion of mismatched donor grafts in the setting of reduced intensity, immune-ablative conditioning for patients with sickle cell disease and other transfusion-dependent anemias should sufficiently achieve engraftment while decreasing the incidence of treatment-related toxicities and achieving an acceptable incidence of graft versus host disease. Utilizing mismatched unrelated volunteer donors and haploidentical related donors will increase the number of patients able to undergo hematopoietic stem cell transplant (HSCT) for these diseases. Additionally, the institutional availability of virus-specific, donor-derived cytotoxic T lymphocytes should address complicated viral infections refractory to standard anti-viral therapy.

The purpose is to:

* To provide alternate donor transplantation from cryopreserved stem cell grafts that are fully characterized for safety and potency to patients with severe sickle cell disease, beta-thalassemia major, or Diamond-Blackfan anemia who do not have matched sibling donor, matched unrelated donor or cord blood donor options.
* To utilize a reduced-intensity conditioning regimen to achieve minimal treatment-related morbidity and mortality while attaining sustained donor engraftment and donor chimerism >20% in order to rescue disease phenotype, specifically in SCD patients.
* To utilize ex-vivo T-cell depletion methods to prevent graft-versus-host disease in the setting of mismatched donor transplantation.
* To utilize additional donor cell products to ensure sufficient immune reconstitution in the immediate post-transplant period, to improve mixed chimerism or provide non-specific anti-viral activity in patients with virus reactivation in the post-transplant period.
* To utilize calcineurin inhibitor-free regimen in an effort to minimize/prevent central nervous system toxicity

ELIGIBILITY:
Inclusion Criteria

1. Patient, parent, or legal guardian must have given written informed consent and/or assent according to FDA guidelines.
2. Ages 5 years to 40 years, at time of consent.
3. Diagnosis of Sickle Cell Disease (Hemoglobin SS, Sβ0-thalassemia) complicated by any of the following:

   * Recurrent acute painful episodes (also known as vaso-occlusive crises; VOC) despite supportive care, minimum of 2 new pain events per year requiring hospitalization for parenteral pain management in the previous 2 years.
   * Recurrent acute chest syndrome (ACS) despite supportive care, minimum of 2 episodes in preceding 2-year period.
   * Stroke or neurologic event lasting > 24 hours with an accompanying infarct on MRI in any patient for all ages; Brain MRI with silent infarct without clinical event in patients ≤ 16 years.
   * Chronic transfusion therapy defined as > 8 packed red blood cell transfusions per year in the year prior to enrollment and/or evidence of red blood cell alloimmunization.
   * Elevated transcranial Doppler velocities - > 200 cm/s, via the non-imaging technique or > 185 cm/s by the imaging technique measured on 2 separate occasions ≥ 1-month apart
   * Elevated TRV > 2.6m/s in patients ≥ 16 years old.
   * Sickle-related renal insufficiency and/or sickle hepatopathy and/or any irreversible end-organ damage in patients ≥ 16 years old.

   OR Diagnosis of beta-thalassemia or Diamond-Blackfan anemia complicated by transfusion dependence with evidence of iron overload.
4. A minimum donor match of 4/8 via high resolution HLA typing at HLA-A, -B, -C, -DRB1 loci in the related setting or minimum donor match of 6/8 via high resolution HLA typing at HLA-A, -B, -C, -DRB1 loci (with the DRB1 locus as a full match requirement). An unrelated donor and cord blood search must have been completed without an eligible 8/8 matched unrelated donor or 6/8 cord blood unit available. Patients who may have acceptable cord blood donor options (4/6 or better) but are limited by cell dose of a single cord will also be eligible for the proposed study.
5. Adequate function of other organ systems as measured by:

   * Creatinine clearance or GFR ≥ 45 ml/min/1.73m.
   * Hepatic transaminases (ALT/AST) ≤ 3 x upper limit of normal.
   * Liver MR imaging for iron content should be performed in all patients with Ferritin > 500 ng/mL. If hepatic iron content > 10mg Fe/g liver should have hepatology consultation and liver biopsy to confirm absence of cirrhosis, fibrosis or hepatitis.
   * Adequate cardiac function as measure by echocardiogram (shortening fraction > 26% or ejection fraction > 40% or >80% of age-specific normal).
   * Pulmonary evaluation testing demonstrating FEV1/FVC ≥ 60% of predicted for age and/or resting pulse oximeter ≥ 92% on room air.
   * Cardiology clearance to proceed with conditioning regimen and HSCT.
   * Pulmonology clearance to proceed with conditioning regimen and HSCT.
6. Subjects must be human immunodeficiency virus (HIV) negative by PCR.
7. Negative pregnancy test for females ≥10 years old or who have reached menarche, unless surgically sterilized.
8. All females of childbearing potential and sexually active males must agree to use an FDA approved method of birth control for up to 24 months after BMT or for as long as they are taking any medication that may harm a pregnancy, an unborn child or may cause a birth defect.
9. Subject and/or parent guardian will also be counseled regarding the potential risks of infertility following BMT and advised to discuss sperm banking or oocyte harvesting (Refer to section,
10. Hydroxyurea must have been trialed and failed in patients with sickle cell disease.

Patient Exclusion Criteria

1. Patients with alternate, superior donor options (matched sibling donor or matched unrelated donor).
2. Patients who have undergone stem cell transplantation in the 6 months prior to anticipated conditioning.
3. Patients with history of a central nervous system (CNS) event within six months prior to start of conditioning (patient will be delayed until eligible).
4. Patients who are pregnant or lactating
5. Patients with uncontrolled bacterial, viral or fungal infection
6. Past or current medical problems or findings from physical examination or laboratory testing that are not listed above, which, in the opinion of the investigator, may pose additional risks from participation in the study, may interfere with the participant's ability to comply with study requirements or that may impact the quality or interpretation of the data obtained from the study.

Ages: 5 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Estimated)
Dates: Start 2018-08-02 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Graft rejection | Day -30 through study completion, an average of 2 years
  How frequent, if any, graft rejection occurs
Post Transplant treatment related mortality | By day 100
  Number of deaths that occurred from treatment
Acute Graft versus host disease | Day 0 through study completion, an average of 2 years
  The number of patients who develop acute graft versus host disease (GVHD)post transplant
Chronic Graft versus host disease | Day 0 through study completion, an average of 2 years
  The number of patients who develop chronic graft versus host disease (GVHD) post transplant
Post Transplant treatment related mortality | Day 180
  Number of deaths that occurred from treatment
Post Transplant treatment related mortality | 1 year
  Number of deaths that occurred from treatment

SECONDARY OUTCOMES:
Neutrophil recovery | Day 0 through study completion, an average of 2 years
  ≥ 0.5 x 103/μL neutrophils for three consecutive days tested on different days.
Donor Cell Engraftment | From Day 0, Day 42, Day 100 and Day 180. Further testing can be done if clinically indicated up to 2 years post transplant
  ≥ 5% donor cells on day +42 and ≥ 10% donor cells on day +100. We will record if subjects have attained robust donor cell engraftment (> 50% donor chimerism at 180 days).
Neurological complications | Day 0 through study completion, an average of 2 years
  To evaluate the incidence of neurological complications
Immune reconstitution | Day 0 through study completion, an average of 2 years
  The pace of systemic immune reconstitution
Cytomegalovirus (CMV) infection | Day 0 through study completion, an average of 2 years
  Incidence of CMV infection by Polymerase chain reaction (PCR) as clinically indicated
Donor Lymphocyte Infusions response | Day 0 through study completion, an average of 2 years
  Evaluate for delayed immune reconstitution, mixed chimerism or viral reactivation
Response to donor-derived virus-specific cytotoxic T-cell therapy | Day 0 through study completion, an average of 2 years
  Activation or reactivation of Cytomegalovirus (CMV), Epstein-Barr Virus (EBV) or adenovirus testing by PCR
Sickle Cell disease phenotype recurrence | Day 0 through study completion, an average of 2 years
  The incidence of Sickle Cell recurrence as clinical evidence of vaso occlusive crisis, detection of HgbS>25% and acute chest syndrome.
Recurrence of transfusion-dependence | Day 0 through study completion, an average of 2 years
  Chronic transfusion therapy defined as > 8 packed red blood cell transfusions per year in the year prior to enrollment and/or evidence of red blood cell alloimmunization.
Organ toxicity | Day 0 through study completion, an average of 2 years
  Incidence of Grade 3-4
Long-term complications-Sterility, endocrinopathy, and secondary malignancy | Day 0 through study completion, an average of 2 years
  Incidence of long term complications
Pediatric Quality of Life Inventory | Baseline through study completion, an average of 2 years
  Measures Pain/Hurt ,Pain Impact,Pain Management/Control ,Worry ,Emotions ,Treatment , Communication
Platelet Recovery | Day 0 through study completion, an average of 2 years
  Platelet count of ≥ 20,000/μL without platelet transfusion in the previous 7 days.
Adult Sickle Cell Quality of Life Measurement System (ASCQ) | Baseline through study completion, an average of 2 years
  Patient reported outcome measurement system that assesses the physical, social and emotional impact of Sickle Cell Disease.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Szabolcs, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No